CLINICAL TRIAL: NCT00364143
Title: A Phase I Study of IHL-305 (Irinotecan Liposome Injection) in Patients With Advanced Solid Tumors
Brief Title: Safety Study of IHL-305 (Irinotecan Liposome Injection) to Treat Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yakult Honsha Co., LTD (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IHL-PRT001
Expanded Access: Available
Record Dates: First submitted 2006-08-11; First posted 2006-08-15 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Cancer
Keywords: Cancer; Advanced Solid Tumor; Oncology
MeSH Terms: conditions — Neoplasms | interventions — irinotecan sucrosofate

INTERVENTIONS:
Drug: IHL-305 (irinotecan liposome injection)

SUMMARY:
The purpose of this study is to determine whether IHL-305 (irinotecan liposome injection) is safe and effective in the treatment of advanced solid tumors.

DETAILED DESCRIPTION:
This is a Phase I dose-escalation study of intravenous administration of IHL-305 in patients with advanced solid tumors. Patients will receive IHL-305 as an intravenous infusion over 60 minutes on Day 1 followed by a 27-day observation period for a total of 28 days (4 weeks) per cycle. Two patient populations will be evaluated separately; patients with UGT1A1*28 genotype homozygous wild-type (wt/wt) and heterozygous (wt/*28) variants as one group, and patients with UGT1A1*28 homozygous variant (*28/*28) as another group.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed malignant solid tumor and not a candidate for known regimens or protocol treatments of higher efficacy or priority
2. Failed conventional therapy for their cancer or have a malignancy for which a conventional therapy does not exist
3. Recovered from all acute adverse effects of prior therapies, excluding alopecia (hair loss)
4. ECOG performance status of 0, 1, or 2
5. 18 years of age or older
6. Normal organ and bone marrow function as defined by:

   * absolute neutrophil count greater than or equal to 1,500 cells/microliter
   * platelets greater than or equal to 100,000 cells/microliter
   * total bilirubin within normal institutional limits
   * AST (SGOT)/ALT (SGPT) less than or equal to 2.5 x institutional upper limit of normal (ULN) or less than or equal to 5.0 x ULN in patients with liver metastases
   * plasma creatinine less than or equal to 1.5 x institutional ULN OR
   * creatinine clearance greater than or equal to 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
7. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

1. Previously treated with irinotecan, or had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study, or not recovered from adverse effects due to agents administered more than 4 weeks earlier
2. Receiving any other investigational agent
3. Known brain metastases
4. History of allergic reactions attributed to compounds of similar chemical composition to IHL-305
5. Concurrent serious infections (i.e., requiring an intravenous antibiotic)
6. Pregnant women or women of childbearing potential and not using methods to avoid pregnancy; a negative pregnancy test (urine or serum) must be documented at baseline for women of childbearing potential; no breast-feeding while on study.
7. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements
8. Significant cardiac disease including heart failure that meets New York Heart Association (NYHA) class III and IV definitions; history of myocardial infarction within one year of study entry; uncontrolled dysrhythmias; or poorly controlled angina.
9. History of serious ventricular arrhythmia (ventricular tachycardia [VT] or ventricular fibrillation [VF], greater than or equal to 3 beats in a row); QTc greater than or equal to 450 msec for men and 470 msec for women; or left ventricular ejection fraction (LVEF) less than or equal to 40% by multi-gated acquisition scan (MUGA).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-09; Study Completion 2011-06

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity within 28 days of treatment administration for patients with UGT1A1*28 genotype (wt/wt and wt/*28)
determination of maximum tolerated dose (MTD) and recommended Phase 2 dose for patients with UGT1A1*28 genotype (wt/wt and wt/*28)

SECONDARY OUTCOMES:
Tumor shrinkage per Response Evaluation Criteria in Solid Tumors (RECIST) every 8 weeks/2 cycles while receiving study drug for patients with UGT1A1*28 genotype (wt/wt and wt/*28)
limited pharmacokinetics (PK) for patients with UGT1A1*28 genotype (wt/wt and wt/*28)
limited incidence and severity of adverse events (AEs) and PK for UGT1A1 homozygous (*28/*28) patients

CONTACTS AND LOCATIONS:
Overall Officials: Mace L Rothenberg, M.D., Principal Investigator — Vanderbilt University
Locations (2):
- United States (2):
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee